CLINICAL TRIAL: NCT03662152
Title: Effects of Vibration Foam Rolling and Non-vibration Foam Rolling in Recovery After Exercise Induce Muscle Damage
Brief Title: Effects of Vibration Foam Rolling After Muscle Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Muñoz-Garcia (Other)
Collaborators: Camilo Jose Cela University (Other)
Responsible Party: Sponsor-Investigator, Daniel Muñoz-Garcia, PhD, Centro Universitario La Salle
Organization: Centro Universitario La Salle (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEI UCJC
Record Dates: First submitted 2018-07-30; First posted 2018-09-07 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Pain, Acute
Keywords: foam roller; vibration foam roller; pressure pain threshold; oxygen saturation; countermovement jump; soreness
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor of data was blinded to statistics investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foam roller (Experimental): Non-Vibration Foam Rolling (NVFR) Group: subjects performed the FR protocol using a custom-made foam roller composed of a polystyrene foam cylinder (15-cm diameter × 35-cm long).
  Interventions: Device: Foam roller
- vibration foam roller (Experimental): Vibration Foam Rolling (VFR) Group: subjects performed the same protocol using a foam roller with vibration (frequency: 18 Hz) composed of a polystyrene foam cylinder (15-cm diameter × 35-cm long) (Hyperice ®).
  Interventions: Device: Vibration foam roller

INTERVENTIONS:
Device: Foam roller — Foam roller massage after DOMS
  Arms: Foam roller
Device: Vibration foam roller — Foam roller massage with vibration after DOMS
  Arms: vibration foam roller

SUMMARY:
Purpose: To compare the effects between non-vibration foam rolling (NVFR) and vibration foam rolling (VFR) on visual analogic scale (VAS), pressure pain threshold (PPT), oxygen saturation (SmO2), counter-movement jump (CMJ), and hip and knee range of movement (ROM) after induction of muscle damage through eccentric acute-exercise using inertial flywheel.

Methods: Thirty-eight healthy subjects (males n=32 females= 6, age 22.2±3.2 years) were randomly assigned in a counter-balanced fashion to either a VFR or NVFR protocol group. All subjects performed a 10x10 (sets x reps) eccentric squat protocol to induce muscle damage. The protocols were administered 48-h post-exercise, measuring VAS, PPT, SmO2, CMJ and ROM, before and immediately post-treatment. The technique of treatment was repeated on both legs for 1 min for a total of 5 sets, with a 30-s rest between sets.

DETAILED DESCRIPTION:
Muscle damage was induced with overload eccentric training using inertial flywheel (2.7-kg flywheels with a moment inertia of 0.07 kg m-2). Immediately after baseline measures, subjects performed 10 sets x 10 repetitions parallel squats using a gravity-free training device flywheel with 2 minutes of recovery between sets. The squat exercise was chosen as basic movement because of its similar muscles recruitment to many athletic movements patterns. Furthermore, the squat exercise is one of the main exercises used to improve the lower-body strength. The required technique was demonstrated to all subjects before beginning the eccentric session, and they were coached during the protocol to be sure adequate technique and maximal effort in each repetition were maintained. All participants performed 5 min on a treadmill to warm up before performing the eccentric bout.

Description of the foam roller intervention The foam-rolling technique was based on a previously published protocol. In both protocols, the technique was repeated on both legs for 1 min for a total of 5 sets, with a 30-s rest between sets. The cadence for both techniques (NVFR and VFR) was fixed at 3:4 using a metronome.

Using a protocol adapted from previous study, subjects began in the plank position with the foam roller at the most proximal portion of the quadriceps of both legs, with as much of their body mass as possible on the foam roller.

Non-Vibration Foam Rolling (NVFR) Group: subjects performed the FR protocol using a custom-made foam roller composed of a polystyrene foam cylinder (15-cm diameter × 35-cm long).

Vibration Foam Rolling (VFR) Group: subjects performed the same protocol using a foam roller with vibration (frequency: 18 Hz) composed of a polystyrene foam cylinder (15-cm diameter × 35-cm long).

ELIGIBILITY:
Inclusion Criteria:

* All subjects were free from musculoskeletal disorders in the last year. All subjects were asked to abstain from unaccustomed exercise, all medications and dietary supplements 72 hours before baseline measurements, during the experimental period and post-treatment

Exclusion Criteria:

* Subjects with symptoms or pathology,

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
visual-analogue scale (VAS) | 2 seconds
  used to measure DOMS and to estimate the intensity of its associated pain. In order to standardize the scaling instructions, the endpoints were described for the subject as 0 = 'no sensation' and 10 = 'the most worst intense sensation imaginable' (16,40). The VAS was measured in four different conditions: 1) passive, 2) during isometric quadriceps contraction, 3) performing a squat and 4) during stretch quadriceps.
Pressure pain threshold | 1 minute
  measured using a digital pressure algometer (Microfet3 ®, Hoggan Health Industries). The digital dynamometer with a 1 cm probe was used to measure three points at the quadriceps: vastus lateralis (VL), rectus femoris (RF) and vastus medialis (VM). Subject was lying on the stretcher, the algometer was positioned perpendicularly to the skin at each point and gradual pressure was applied until the subject reported a change from the sensation of pressure to pain. In that point the pressure was stopped immediately and the value was recorded represented the pain threshold (16). The mean of the 3 measures was calculated. Algometry has been shown to be highly reliable (ICC = 0.91) (9).
Muscle oxygenation | 2 minutes
  was recorded at rest, during 10 squat repetitions (body weight load) and immediately after, using a commercially available portable non-invasive near infrared spectroscopy (NIRS) device (Moxy, Fortiori Design LLC, Minnesota, USA).

SECONDARY OUTCOMES:
Infrared Optojump photoelectric cells (Microgate Corporation, Bolzano, Italy) | 5 minutes
  were used to measure explosive strength in lower limbs
Passive and active hip extension and knee flexion ROM of the dominant leg | 2 minutes
  were measured with a Microfet3 ® inclinometer using the protocol of Norkin & White

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Superior de Estudios Universitarios La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No